CLINICAL TRIAL: NCT03361735
Title: A Phase 2 Trial of Radium Ra 223 Dichloride in Combination With Androgen Deprivation Therapy and Stereotactic Body Radiation Therapy for Patients With Oligometastatic Castration Sensitive Prostate Cancer
Brief Title: Radium Ra 223 Dichloride, Hormone Therapy and Stereotactic Body Radiation Therapy in Treating Patients With Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17085; NCI-2017-02192 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma
Keywords: PSA Level Greater than or Equal to 0.2; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Leuprolide; luprolide acetate gel depot; Goserelin; Radiosurgery; radium Ra 223 dichloride; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (hormone therapy, SBRT, radium Ra 223 dichloride) (Experimental): Beginning 4 weeks (28 days) prior to radiation therapy, patients receive leuprolide acetate or goserelin acetate, for up to 32 weeks. Patients also undergo 3-5 fractions of SBRT every 40 hours over 7-21 days beginning on day 1 of course 1, and receive radium Ra 223 dichloride IV over 1 minute on day 1 of courses 2-7. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Radiation: Stereotactic Body Radiation Therapy; Radiation: Radium Ra 223 Dichloride; Other: Laboratory Biomarker Analysis; Drug: Degarelix

INTERVENTIONS:
Drug: Leuprolide Acetate — Intramuscular or subcutaneous injection
  Other Names: 377526; 6-D-Leucine-9-(N-ethyl-L-prolinamide)-1-9-luteinizing Hormone-releasing Factor (Pig) Monoacetate; 6-D-Leucine-9-(N-ethyl-L-prolinamide)-10-deglycinamide Luteinizing Hormone-Releasing Factor (Pig) Monoacetate; 74381-53-6; A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Goserelin Acetate — Subcutaneous injection
  Other Names: 606864; 65807-02-5; D-Ser(bu(t))(6)azgly(10)-LHRH Acetate; ZDX; Zoladex
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: 444811-40-9; Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM CHLORIDE RA-223; Radium-223 Dichloride; Xofigo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Degarelix — Subcutaneous injection
  Other Names: 214766-78-6; FE200486; Firmagon

SUMMARY:
This phase 2 trial studies radium Ra 223 dichloride, hormone therapy and stereotactic body radiation in treating patients with prostate cancer that has spread to other places in the body. Radium Ra 223 dichloride contains a radioactive substance that collects in the bone and gives off radiation that may kill cancer cells. Hormone therapy using leuprolide acetate or goserelin acetate may fight prostate cancer by lowering the amount of testosterone the body makes. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Giving radium Ra 223 dichloride, hormone therapy and stereotactic body radiation may work better at treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the time to treatment failure (TTF) in patients who initiated the protocol regimen of androgen deprivation therapy (ADT) with stereotactic body radiation therapy (SBRT) and radium Ra 223 dichloride and received at least one dose with radium Ra 223 dichloride.

SECONDARY OBJECTIVES:

I. To assess the safety of adding radium Ra 223 dichloride to SBRT and ADT in patients with oligometastatic castration sensitive prostate cancer.

II. To assess the prostate-specific antigen (PSA) and overall response rate (ORR) after 6 cycles of radium Ra 223 dichloride (cycle 8 day 1).

III. To assess the progression-free survival (PFS) in patients with oligometastatic castration sensitive prostate cancer who initiated the protocol regimen of ADT with SBRT and radium Ra 223 dichloride and received at least one dose of radium Ra 223 dichloride.

IV. To assess time to bone specific PFS in patients with oligometastatic castration sensitive prostate cancer who initiated the protocol regimen of ADT with SBRT and radium Ra 223 dichloride and received at least one dose of radium Ra 223 dichloride.

V. To assess overall survival, complete response rate, duration of response, and duration of overall complete response and duration of stable disease in patients with oligometastatic castration sensitive prostate cancer who initiated the protocol regimen of ADT with SBRT and radium Ra 223 dichloride.

VI. To assess long-term toxicities during 5-year follow-up in patients with oligometastatic castration sensitive prostate cancer who initiated the protocol regimen of ADT with SBRT and radium Ra 223 dichloride and received at least one dose of radium Ra 223 dichloride.

TERTIARY OBJECTIVES:

I. To perform exploratory analysis of primary or metastatic tumor mutation patterns in this study population at baseline.

II. To identify immune system factors in the blood that change during the course of ADT-radiotherapy for metastatic prostate cancer.

III. To describe the rate of normalization of the total alkaline phosphatase level (defined as a return to a value within the normal range) at the end of protocol therapy in patients oligometastatic castration sensitive prostate cancer with total alkaline phosphatase values above the upper limit of the normal range at baseline.

OUTLINE:

Beginning 4 weeks (28 days) prior to radiation therapy, patients receive leuprolide acetate or goserelin acetate, or degarelix for up to 32 weeks. Patients also undergo 3-5 fractions of SBRT every 40 hours over 7-21 days beginning on day 1 of course 1, and receive radium Ra 223 dichloride intravenously (IV) over 1 minute on day 1 of courses 2-7. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of participant and/or legally authorized representative
* Agreement to provide archival primary or metastatic tumor tissue if available
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Life expectancy > 12 months
* Histologic diagnosis of prostate adenocarcinoma

  * Pure small cell carcinoma will be excluded; however, component of neuroendocrine /small cell differentiation will be allowed provided that adenocarcinoma constitutes majority of the tissue specimen
* Stage M1

  * Metastatic disease can be documented by bone scan or computed tomography (CT) scan or magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT or the combination of these tests
* Up to 4 metastatic lesions:

  * Must have at least 1 bone lesion AND each non-visceral lesion should be less than 5 cm
  * Visceral lesions will be limited to one lung lesion (< 2 cm) or one lymph node; no liver lesions allowed; lymph nodes allowed provided they are not in a field of prior radiation, and if amenable to SBRT (to be reviewed by principal investigator [PI])
* Two lesions can be in close proximity (i.e. within 5 cm of each other) if they meet radiation SBRT normal tissue toxicity requirements
* If have untreated primary prostate cancer: must undergo debulking prostatectomy
* If had prior definitive radiation therapy to the prostate: no evidence of locally persistent or recurrent prostate cancer on digital rectal exam (DRE) and imaging studies (CT or MRI); retreatment to local residual-recurrent disease will result in potential eligibility to be reviewed by PI on a case-by-case basis
* Does not have castration resistant disease

  * Castration resistance defined as progression of disease despite serum testosterone level of < 50 ng/dL
* PSA >= 0.2 prior to start of androgen deprivation treatment
* Initiated 28 (+ 7) days of androgen deprivation therapy (ADT) prior to day 1 of protocol therapy

  * Only luteinizing hormone-releasing hormone (LHRH) agonist/antagonist treatment is considered ADT, bicalutamide or other antiandrogens used alone do not count
* May have received prior hormonal therapy in the context of definitive treatment of a primary tumor

  * Patients may have had one prior systemic non-chemotherapeutic treatment (i.e. immunotherapy, receptor tyrosine kinase inhibitor, antiangiogenic agent, differentiating agent) for recurrent or metastatic disease
* Must have refused standard of care chemotherapy for metastatic disease
* Recovered from all acute side-effects (except alopecia) related to previous systemic therapy
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (to be performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: growth factor support is not permitted to normalize baseline ANC parameters, however subsequent growth factor administration is permitted as standard supportive care
* Platelets >= 100,000/mm^3 (to be performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: transfusion of blood products are not allowed to normalize baseline blood parameters, however subsequent transfusions are allowed per standard supportive care guidelines
* Hemoglobin (HgB) >= 9.0 g/dL (to be performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: transfusion of blood products are not allowed to normalize baseline blood parameters, however subsequent transfusions are allowed per standard supportive care guidelines
* Total serum bilirubin =< 2 x upper limit of normal (ULN) (to be performed within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (to be performed within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (to be performed within 14 days prior to day 1 of protocol therapy)
* Creatinine =< 2.5 mg/dL (to be performed within 14 days prior to day 1 of protocol therapy)

Exclusion Criteria:

* Prior radium Ra 223 dichloride
* Prior or concomitant chemotherapy for metastatic or recurrent disease with the following exceptions:

  * Prior chemotherapy for local primary disease is permitted
  * Bisphosphonates or receptor activator of nuclear factor kappa-Β (RANK) ligand inhibitors are allowed at doses and schedule consistent with the treatment or prevention of osteoporosis
* Prior radiation treatment for metastatic disease
* Concomitant radiation treatment to primary prostate site
* Orchiectomy
* Unstable medical comorbidities (i.e. uncontrolled cardiac comorbidities)
* Metastases that in the judgment of investigator-radiologist are not amenable to SBRT
* History of brain metastases or who currently have treated or untreated brain metastases
* Uncontrolled human immunodeficiency virus (HIV) infection
* Any other condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | Assessed up to 5 years
  Defined as time from the initiation of androgen deprivation therapy (ADT) for metastatic disease until PSA increase to > pre-ADT level or PSA > 10 (whichever is smaller) or radiographic or clinical progression or resumption of ADT by physician's choice.
Objective response rate | Up to 5 years
  Response will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria. Proportion of patients achieving complete response (CR) or partial response (PR) at course 8, day 1 (post 6 doses of radium Ra 223 dichloride).

SECONDARY OUTCOMES:
Progression-free survival | From the initiation of ADT for metastatic disease until PSA progression or radiographic progression or death, assessed up to 5 years
  Progression will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Overall survival | From date of initiation of protocol treatment to date of death from any cause, assessed up to 5 years
Complete response (CR) rate defined as the proportion of patients achieving CR | Up to 5 years
  Response will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Duration of response | From documented response to recurrent or progressive disease is first met, assessed up to 5 years
  Response will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Duration of overall complete response | From documented CR to recurrent/ progressive disease, assessed up to 5 years
  Response will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Bone specific progression-free survival | Time to progression of bone specific disease over baseline, assessed up to 5 years
  Progression will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Duration of stable disease | Time from start of treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, assessed up to 5 years
  Response will be evaluated in this study using modified Prostate Cancer Working Group 2 criteria.
Incidence of adverse events (AE) graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years
  Toxicity will be graded. The highest AE grade per cycle will be reported in the electronic case report form (eCRF) from start of therapy until the end of treatment visit.

OTHER OUTCOMES:
Rate of normalization of the total alkaline phosphatase level | Baseline up to 5 years
  The rate of normalization of the total alkaline phosphatase level (defined as a return to a value within the normal range) at the end of protocol therapy in patients with total alkaline phosphatase values above the upper limit of the normal range at baseline will be assessed.
Genomic mutations analysis | Up to 5 years
Immune biomarker analysis | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Savita Dandapani, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States